CLINICAL TRIAL: NCT00114361
Title: Peginterferon Alfa-2a and Ribavirin Combination Therapy in Patients With HBeAg-negative Chronic HBV Infection (PARC Study)
Brief Title: 48 Weeks Combination Therapy for Patients With HBeAg-negative Chronic Hepatitis B Virus (HBV) Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Foundation for Liver Research (Other)
Responsible Party: Prof. H.L.A. Janssen, Foundation for Liver reseach
Allocation: Randomized | Model: Factorial | Masking: Double
Other Study IDs: HBV05-01; EudraCT: 2004-004736-30
Record Dates: First submitted 2005-06-14; First posted 2005-06-15 (Estimated); Last update posted 2010-06-22 (Estimated); Status verified 2010-06

CONDITIONS: Hepatitis B
Keywords: HBeAg-negative; chronic; hepatitis B; viral
MeSH Terms: conditions — Hepatitis B; Bronchiolitis Obliterans Syndrome | interventions — Ribavirin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Ribavirin + Peg IFN
  Interventions: Drug: Ribavirin
- 2 (Active Comparator): Peg IFN + Placebo
  Interventions: Drug: Peginterferon alpha 2a

INTERVENTIONS:
Drug: Ribavirin — 1200 mg a day, 48 weeks
  Arms: 1
Drug: Peginterferon alpha 2a — 180 µg per week, 48 weeks
  Arms: 2

SUMMARY:
The purpose of this study is to investigate whether in patients with chronic HBeAg-negative hepatitis B, PEG-IFN-ribavirin combination therapy for 1 year leads to enhanced response (HBV DNA <10E4 copies/ml and normal ALT 24 weeks after treatment discontinuation) in comparison with pegylated interferon (PEG-IFN) monotherapy.

DETAILED DESCRIPTION:
Despite the introduction of newer drugs for the treatment of chronic hepatitis B, there is still no optimal treatment. Pegylated interferon alfa has proven sustained efficacy in approximately 30-40% of patients with HBeAg-positive or HBeAg-negative chronic hepatitis B. It is likely that combination therapy of pegylated interferon alfa with ribavirin in chronic hepatitis B is more effective than pegylated interferon alfa monotherapy. In chronic hepatitis C, adding ribavirin to pegylated interferon therapy doubled the sustained response rate (29% vs. 56%) and has become the standard option of treatment.

To investigate the effect of the treatment with pegylated interferon and ribavirin on the amount of inflammation and fibrosis in the liver, a liver biopsy will be performed within one year prior to screening and at the end of follow-up.

When patients with chronic hepatitis B are treated outside any study with pegylated interferon, they visit the outpatient clinic approximately every month for blood samples. So in this study the amount of blood samples taken from every patient is not increased as compared with treatment outside a study.

ELIGIBILITY:
Inclusion Criteria:

* Chronic hepatitis B
* Biopsy performed within one year prior to screening or during screening
* ALT > 1.5 x ULN
* HBeAg negative, anti-HBeAg positive
* HBV DNA > 10E5 copies/ml
* Age 18-70 years
* Written informed consent
* Hepatic imaging without evidence of HCC
* All fertile males and females must be using two forms of effective contraception

Exclusion Criteria:

* Antiviral therapy against HBV within the previous 6 months; treatment with any investigational drug within 30 days of entry to this protocol
* Severe hepatitis activity as documented by ALT > 10 x ULN
* Advanced liver disease
* Pre-existent leucopenia or thrombopenia
* Co-infection with HCV,HDV or HIV
* Other acquired or inherited causes of liver disease
* Alpha fetoprotein > 50 ng/ml.
* Evidence of severe renal disease
* Hyper- or hypothyroidism
* Significant cardiovascular or pulmonary dysfunction, malignancy,immunodeficiency syndromes
* Immune suppressive treatment within the previous 6 months
* Contra-indications for alpha-interferon therapy
* Pregnancy, breast-feeding
* Any medical condition requiring chronic systemic administration of steroids
* Substance alcohol or drug abuse
* Subjects with clinically significant retinal abnormalities
* Subjects with clinically significant hearing abnormalities
* Hemoglobinopathies
* Subjects with known hypersensitivity to ribavirin

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2005-03; Primary Completion 2008-05 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
The combined presence of HBV DNA level < 10E4 copies/ml and ALT normalization at the end of follow-up | may 2008

SECONDARY OUTCOMES:
ALT normalization | May 2008
HBV DNA negativity(undetectable by Taqman PCR) | May 2008
HBsAg loss from serum | May 2008
Improvement liver histology | May 2008
Combined virological, biochemical and histological response | May 2008

CONTACTS AND LOCATIONS:
Overall Officials: Harry LA Janssen, MD PhD, Principal Investigator — Foundation of Liver Research
Locations (1):
- Erasmus MC department hepatology, Rotterdam, Netherlands

REFERENCES:
- [Derived] Brakenhoff SM, de Knegt RJ, van Campenhout MJH, van der Eijk AA, Brouwer WP, van Bommel F, Boonstra A, Hansen BE, Berg T, Janssen HLA, de Man RA, Sonneveld MJ. End-of-treatment HBsAg, HBcrAg and HBV RNA predict the risk of off-treatment ALT flares in chronic hepatitis B patients. J Microbiol Immunol Infect. 2023 Feb;56(1):31-39. doi: 10.1016/j.jmii.2022.06.002. Epub 2022 Jul 2. PMID 35941076
- [Derived] Brakenhoff SM, de Knegt RJ, Oliveira J, van der Eijk AA, van Vuuren AJ, Hansen BE, Janssen HLA, de Man RA, Boonstra A, Sonneveld MJ. Levels of Antibodies to Hepatitis B Core Antigen Are Associated With Liver Inflammation and Response to Peginterferon in Patients With Chronic Hepatitis B. J Infect Dis. 2022 Dec 28;227(1):113-122. doi: 10.1093/infdis/jiac210. PMID 35599306
- [Derived] Brakenhoff SM, de Man RA, Boonstra A, van Campenhout MJH, de Knegt RJ, van Bommel F, van der Eijk AA, Berg T, Hansen BE, Janssen HLA, Sonneveld MJ. Hepatitis B virus RNA decline without concomitant viral antigen decrease is associated with a low probability of sustained response and hepatitis B surface antigen loss. Aliment Pharmacol Ther. 2021 Jan;53(2):314-320. doi: 10.1111/apt.16172. Epub 2020 Nov 21. PMID 33222190
- [Derived] Farag MS, van Campenhout MJH, Pfefferkorn M, Fischer J, Deichsel D, Boonstra A, van Vuuren AJ, Ferenci P, Feld JJ, Berg T, Hansen BE, van Bommel F, Janssen HLA. Hepatitis B Virus RNA as Early Predictor for Response to Pegylated Interferon Alpha in HBeAg-Negative Chronic Hepatitis B. Clin Infect Dis. 2021 Jan 27;72(2):202-211. doi: 10.1093/cid/ciaa013. PMID 31912157